CLINICAL TRIAL: NCT03880682
Title: Treatment of Chronic Hepatitis C Virus Infection With Direct Acting Antivirals in Kidney Transplant Recipients
Brief Title: Direct Acting Antivirals for HCV Infection in Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Safak Mirioglu, Principal Investigator, Istanbul University
Other Study IDs: 2018/1511
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Kidney Transplant; Complications; Hepatitis C, Chronic
Keywords: kidney transplant recipients; chronic hepatitis c virus infection; direct acting antivirals; sofosbuvir/ledipasvir
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Kidney transplant recipients with chronic HCV infection who were treated using direct acting antivirals.

SUMMARY:
Chronic hepatitis C virus (HCV) infection, an important cause of morbidity and mortality worldwide, is a significant problem in kidney transplant recipients (KTRs) given its high prevalence in patients undergoing hemodialysis. Interferon based regimens were cornerstone of treatment of HCV infection in the past; however, due to their low efficacy and high rates of adverse effects, they have been abandoned in the new era of direct acting antivirals (DAAs). Several studies demonstrated the efficacy and safety of DAAs, yet data regarding clinical practice of these agents in KTRs is still needed. Therefore, we conducted a study using our registry data to evaluate the efficacy and safety of DAAs in KTRs.

ELIGIBILITY:
Inclusion Criteria:

* Being a kidney transplant recipient.
* Having a detectable level of HCV RNA.
* Having direct acting antivirals for 12 or 24 weeks.

Exclusion Criteria:

* Withdrawing or not providing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients with chronic HCV infection who were treated using direct acting antivirals.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
SVR12 | 6 months
  Undetectable levels of HCV RNA for 12 weeks after the end of treatment with direct acting antivirals.

SECONDARY OUTCOMES:
Stable Graft Function | 6-12 months
  Stability of serum creatinine and proteinuria levels of kidney transplant recipients during and after the treatment with direct acting antivirals.
Stable Serum Trough Levels of Immunosuppressive Agents | 6 months
  Stability of serum trough levels of calcineurin and mTOR inhibitors during the treatment with direct acting antivirals.

CONTACTS AND LOCATIONS:
Overall Officials: Safak Mirioglu, MD, Principal Investigator — Department of Internal Medicine, Istanbul Faculty of Medicine; Halil Yazici, MD, Study Chair — Department of Internal Medicine, Istanbul Faculty of Medicine; Sabahattin Kaymakoglu, MD, Study Chair — Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colombo M, Aghemo A, Liu H, Zhang J, Dvory-Sobol H, Hyland R, Yun C, Massetto B, Brainard DM, McHutchison JG, Bourliere M, Peck-Radosavljevic M, Manns M, Pol S. Treatment With Ledipasvir-Sofosbuvir for 12 or 24 Weeks in Kidney Transplant Recipients With Chronic Hepatitis C Virus Genotype 1 or 4 Infection: A Randomized Trial. Ann Intern Med. 2017 Jan 17;166(2):109-117. doi: 10.7326/M16-1205. Epub 2016 Nov 15. PMID 27842383